CLINICAL TRIAL: NCT05444686
Title: Comparative Study of 99mTc-FAPI Quantitative SPECT/CT and 68Ga-FAPI PET/CT in Clinical Diagnosis and Staging of Gastrointestinal Tumors
Brief Title: Comparative Study of 99mTc-FAPI SPECT/CT and 68Ga-FAPI PET/CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20222134-C
Record Dates: First submitted 2022-06-26; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: 99mTc-FAPI-positive Gastrointestinal Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 99mTc-FAPI — inject the tracer to subjects and perform SPECT/CT scans

SUMMARY:
The purpose of this study is to compare the similarities and differences of 99mTc-FAPI quantitative SPECT/CT and 68Ga-FAPI PET/CT in the diagnosis and staging of gastrointestinal tumors, and clinical diagnosis and economic value of 99mTc-FAPI quantitative SPECT/CT for the gastrointestinal tumors.

DETAILED DESCRIPTION:
5 healthy volunteers with whole body 99mTc-FAPI quantitative SPECT/CT scans at 1, 2, 4, 6 and 24 hours after tracer injection (mean dose, 20.0 ± 2.0 mCi) will be performed. During the imaging period, 1 mL blood samples will be obtained specifically at 1, 2, 4, 6 and 24 hours after the injection, for time-activity curve calculations. The estimated radiation doses will be calculated by using OLINDA/EXM software.

Forty patients with confirmed or suspected gastrointestinal tumors, whole body 99mTc-FAPI quantitative SPECT/CT scans will be performed on the first day, and whole body 68Ga-FAPI PET/CT scans will be performed on the next day.According to the scans results of the two agents, with SUVmax and SUVmean as the analysis indicators, the number and uptake difference of primary tumor and metastatic lesions will be compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients with gastrointestinal tumors: diagnosed by pathological needle biopsy

Exclusion Criteria:

* refuse or cannot endure surgery pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
SUV of primary and metastases lesions | 2 hours after injection
  The standardized uptake values (SUV) in deferent organs and lesions

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruan Q, Zhou C, Wang Q, Kang F, Jiang Y, Li G, Feng J, Zong S, Zhang J, Wang J. A Simple Kit Formulation for Preparation and Exploratory Human Studies of a Novel 99mTc-Labeled Fibroblast Activation Protein Inhibitor Tracer for Imaging of the Fibroblast Activation Protein in Cancers. Mol Pharm. 2023 Jun 5;20(6):2942-2950. doi: 10.1021/acs.molpharmaceut.2c01094. Epub 2023 Apr 21. PMID 37083360